CLINICAL TRIAL: NCT05351437
Title: A Phase l, Single-blind, Placebo-controlled Trial Designed to Assess the Safety and Tolerability of a Single Intravenous Dose of MTx-COVAB36 in Healthy Volunteers.
Brief Title: To Assess the Safety and Tolerability of MTx-COVAB36 as a Therapeutic and Prophylactic Treatment Against COVID-19.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memo Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MTx-COVAB36-AU-1.02CoV
Record Dates: First submitted 2022-03-28; First posted 2022-04-28 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: SARS-CoV-2 Infection
MeSH Terms: conditions — COVID-19 | interventions — MTX-COVAB36

STUDY DESIGN:
Intervention Model Description: Single-blind, placebo-controlled study in healthy volunteers. The trial will comprise four dose cohorts, each composed of 6 participants receiving MTx-COVAB36 and 2 participants receiving placebo, with pre-defined dose levels.
  The predefined investigational medicinal product (IMP) doses are: 100 mg, 500 mg, 1,000 mg and 2,000 mg, respectively. Participants will be randomized into study arms (MTx-COVAB36 or placebo).
Who Masked: Participant
Masking Description: Single-blind study where participants are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTx-COVAB36 (Active Comparator): Cohort 1 - 100 mg IV dose Cohort 2 - 500 mg IV dose Cohort 3 - 1000 mg IV dose Cohort 4 - 2000 mg IV dose MTx-COVAB36 will be administered as a single dose intravenously.
  Interventions: Drug: MTx-COVAB36
- Placebo (Placebo Comparator): Placebo (0.9% NaCl) will be administered as a single dose intravenously.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MTx-COVAB36 — MTx-COVAB36 is a fully human monoclonal IgG1 antibody derived from the memory B cells of convalescent COVID-19 donors and directed against SARS-CoV-2 spike protein with potent virus neutralising activity.
  Arms: MTx-COVAB36
Drug: Placebo — 0.9% saline
  Arms: Placebo

SUMMARY:
This is a single blind, placebo-controlled clinical trial designed to determine the safety and tolerability of MTx-COVAB36 after a single administration in a dose escalation, dose limiting toxicity (DLT)-driven approach in healthy volunteers. Additional data to define the recommended phase II dose (RP2D) will also be determined.

MTx-COVAB36 is a fully human monoclonal IgG1 antibody derived from the memory B cells of convalescent COVID-19 donors and directed against SARS-CoV-2 spike protein with potent virus neutralising activity.

The trial will comprise four dose cohorts, each composed of 6 participants receiving MTx-COVAB36 and 2 participants receiving placebo, with pre-defined dose levels. The pre-defined investigational medicinal product (IMP) doses are: 100 mg, 500 mg, 1,000 mg and 2,000 mg, respectively. Participants will be administered a single dose of either IMP or placebo on Day 1 of the study and will be followed up until 63 days post administration.

DETAILED DESCRIPTION:
Despite the rapid rollout of vaccines against the Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), there is still a need for therapeutic and prophylactic treatments against the Coronavirus Disease 2019 (COVID-19) especially for those individuals who are not sufficiently protected by vaccines, i.e., a significant proportion of people of older age, the immunocompromised and those having various comorbidities.

MTx-COVAB36 is a fully human monoclonal IgG1 antibody derived from the memory B cells of convalescent COVID-19 donors and directed against SARS-CoV-2 spike protein with potent virus neutralising activity.

This is a single blind, placebo-controlled clinical trial designed to determine the safety and tolerability of MTx-COVAB36 after a single administration in a dose escalation, DLT-driven approach in healthy volunteers. Additional data to define the RP2D will also be determined.

The trial will comprise four dose cohorts, each composed of 6 participants receiving MTx-COVAB36 and 2 participants receiving placebo, with pre-defined dose levels. The pre-defined IMP doses are: 100 mg, 500 mg, 1,000 mg and 2,000 mg, respectively. Participants will be administered a single dose of either IMP or placebo on Day 1 of the study and will be followed up until 63 days post administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants aged 18 years to 50 years at the time of consent
2. Ability to read, understand and provide written informed consent
3. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
4. Healthy participants as established by medical history, laboratory examination, physical examination, vital signs, and ECG during screening and as per the clinical judgment of the investigator
5. Body mass index (BMI) 18.0 to 32.0 kg/m2 (inclusive)
6. For Woman of Childbearing Potential (WOCBP): agrees to practice true abstinence or agrees to use a highly effective method of contraception consistently from 30 days prior to Day 1 until end of the study (Day 63). Highly effective contraception includes hormonal contraception, placement of intrauterine device (IUD) or intrauterine system (IUS), or a vasectomized partner (performed at least 6 months prior to her screening) who has been documented to no longer produce sperm. Verbal confirmation from the participant through medical interview is acceptable. No contraception requirements for participants in exclusive same-sex relationship.
7. For male participant: must agree to practice true abstinence or use condom if he has a partner of childbearing potential, or must be surgically sterilized (performed at least 6 months prior and documented to no longer produce sperm. Verbal confirmation through medical nterview is acceptable). Participant to practice abstinence (if applicable) or use condom until end of the study (Day 63). No contraception requirements for participants in exclusive same-sex relationship.
8. Accessible veins in the forearms for venepuncture and/or intravenous cannulation

Exclusion Criteria:

1. Participant with active SARS-CoV-2 infection, verified by RT-PCR test
2. Participants tested positive for human immunodeficiency virus (HIV antibody screen), Hepatitis B virus (HBsAg screen) or Hepatitis C virus (HCV antibody screen)
3. History of administration of any investigational or non-registered drug within 30 days or 5 half-lives, whichever is longer, prior to administration of study drug, or planned administration during the course of study participation
4. History of any reaction to monoclonal antibodies
5. History of clinically relevant atopic diseases and/or known allergies to the trial product or its components
6. History of any major pulmonary, cardiovascular, renal, neurological (e.g., cerebrovascular events), metabolic, gastrointestinal, hepato-biliary, or hematological functional abnormality, malignancy (except for adequately treated basal cell carcinoma or squamous cell carcinoma of the skin), or mental disability as per discretion of the investigator
7. Any clinically significant laboratory findings at screening and enrolment and at Day-1; one retest is allowed at screening and/or at Day-1
8. Acute illness (moderate or severe) and/or fever (body temperature ≥ 38 °C) during the 72 hours prior to planned study drug application
9. Participants with altered immunocompetence such as participants with ongoing cancer treatment, human immunodeficiency virus infection, organ transplant or any other active immune system disorder
10. Receipt of immunoglobulin or blood products within 6 months prior to enrolment
11. Receipt of a monoclonal antibody within previous 6 months or 5 half-lives, whichever is longer
12. Planned surgery (excluding minor procedures such as tooth extraction or incision and drainage) during the course of the study
13. Receipt of any standard vaccine within 14 days prior to Day 1
14. History of alcoholism or drug addiction (as per DSM-V) within 1 year prior to screening
15. Use of prescription drugs within 7 days prior to Day 1 or for 5 half-lives whichever is longer, or during the study, except for hormonal contraceptives or positive result in urine drug screen or alcohol breath test at screening or Day-1
16. Use of over-the-counter medication within 7 days prior to Day 1 or during the study; medication such as paracetamol and ibuprofen may be permitted at the discretion of the investigator and sponsor
17. Receipt of immunosuppressive medications within 6 months prior to enrolment, or any active or prior history of immunodeficiency (receipt of any course of systemic corticosteroids for more than a 7-day duration and with a prednisolone equivalent dose of more than 5 mg per day within 6 months prior to enrolment will exclude a participant; inhaled or topical steroids are allowed)
18. Pregnant, lactating, or planned pregnancy during the study period
19. Inability to comply with the study protocol in the opinion of the investigator
20. Participant has any plans to permanently relocate from the area prior to the completion of the study or to leave for an extended period of time when study visits would need to be scheduled
21. Concurrent participation in another interventional clinical study investigating a vaccine, drug, medical device, or medical procedure in the 30 days preceding the study drug administration or during the course of the study
22. Abnormal vital signs including systolic blood pressure (SBP) < 90 or > 150 mmHg, diastolic blood pressure (DBP) < 40 or > 90 mmHg, heart rate (HR) < 40 or > 100 bpm (average of triplicate measurements) at screening

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2022-09-04 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Day 1 (IMP administration day) to Day 63 (Final visit)
  To investigate the incidence, severity and causal relationship of AEs following single dose IV administration of MTx-COVAB36 to healthy volunteers.

SECONDARY OUTCOMES:
Pharmacokinetics measured by the maximum plasma concentration (Cmax) | Day 1 (IMP administration day) to Day 63 (Final visit)
  To describe the pharmacokinetics of MTx-COVAB36 in healthy volunteers after single dose intravenous administration.
Pharmacokinetics measured by the area under the concentration-time curve (AUC) | Day 1 (IMP administration day) to Day 63 (Final visit)
  To describe the pharmacokinetics of MTx-COVAB36 in healthy volunteers after single dose intravenous administration.
Pharmacokinetics measured by the apparent clearance (CL) | Day 1 (IMP administration day) to Day 63 (Final visit)
  To describe the pharmacokinetics of MTx-COVAB36 in healthy volunteers after single dose intravenous administration.
Pharmacokinetics measured by the terminal half-life (t1/2) | Day 1 (IMP administration day) to Day 63 (Final visit)
  To describe the pharmacokinetics of MTx-COVAB36 in healthy volunteers after single dose intravenous administration.
Immunogenicity measured by anti-drug antibody (ADA) production | Day 1 (IMP administration day), Day 8 and Day 29 post-administration and at Day 63 (final visit).
  Assessment of the incidence and intensity of ADA production
Immunogenicity measured by drug neutralizing antibody (Nab) production | Day 1 (IMP administration day), Day 8 and Day 29 post-administration and at Day 63 (final visit).
  Assessment of the incidence and intensity of Nab production.

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No
The Sponsor, will not be sharing data with anyone outside of Vakzine Projekt Management (VPM GmbH) and the CRO (Accelagen) involved in the study.